CLINICAL TRIAL: NCT06627335
Title: Pregnancy Outcomes Study of Women With Atopic Dermatitis Exposed to Ruxolitinib Cream Versus Topical Corticosteroids During Pregnancy: A US Claims Database Analysis
Brief Title: An Observational Retrospective Cohort Study Being Conducted in Women With Atopic Dermatitis Exposed to Ruxolitinib Cream Versus Topical Corticosteroids During Pregnancy: A US Claims Database Analysis
Status: Recruiting | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB18424-MA-IAI-403
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Atopic Dermatitis
Keywords: ruxolitinib; Atopic Dermatitis; pruritus; eczema; topical therapy; JAK inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants of women with AD exposed to ruxolitinib cream during pregnancy
  Interventions: Drug: Ruxolitinib Cream
- Infants of women with AD exposed to a TCS prior to or during pregnancy
  Interventions: Drug: TCS

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib Cream
  Other Names: Opzelura
  Groups: Infants of women with AD exposed to ruxolitinib cream during pregnancy
Drug: TCS — Topical corticosteroid
  Groups: Infants of women with AD exposed to a TCS prior to or during pregnancy

SUMMARY:
This study is to assess infant outcomes of women with AD who were exposed to ruxolitinib cream during pregnancy compared with a control cohort of women with AD who were exposed to a topical corticosteroid (TCS) during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 14 years or older at pregnancy outcome.
* Pregnancy following FDA approval of ruxolitinib cream for AD on 21 SEP 2021.
* At least 1 pharmacy-dispensing claim for ruxolitinib cream (ruxolitinib-exposed cohort) or a TCS (TCS-exposed cohort).
* A diagnosis of AD prior to or on the day of the first pharmacy claim for ruxolitinib cream (ruxolitinib-exposed cohort) or a TCS (TCS-exposed cohort) from 6 months before the estimated date of conception.
* Continuous enrollment in the database from 6 months before the estimated date of conception through the end of pregnancy.
* For infant outcomes only, linkage of mother and infant data will be required (ie, pregnancies that cannot be linked to an infant will be excluded for infant outcomes but not for pregnancy outcomes). Infants will be followed for as long as they are continuously enrolled in the database up to 1 year after birth (ie, variable follow-up for each infant). A 1-year fixed period of continuous enrollment after birth will not be imposed so as not to introduce survival bias.

Exclusion Criteria:

• One or more pharmacy claims for oral ruxolitinib or other JAK inhibitors in the exposure window for a given outcome.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Exposure cohort study of women within the US with atopic dermatitis (AD) who were exposed to ruxolitinib cream at any time during their pregnancy period.
Sampling Method: Non-Probability Sample
Enrollment: 5621 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of major congenital malformation (MCM)s | Up to 12 months after birth
  Defined as any major structural or chromosomal defect in live-born infants, stillbirths or spontaneous losses equal to or greater than 20 weeks' gestation, or electively terminated pregnancies of any gestational age.

SECONDARY OUTCOMES:
Number of small-for-gestational age (SGA) births | At time of delivery
  Defined as a birthweight at or below the 10th percentile for a given gestational age.
Number of Pregnancy outcomes | Up to birth
  Number of live births, still births, recognized spontaneous abortions and number of elective terminations as defined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Syneos Health (remote site), Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: An Observational Retrospective Cohort Study Being Conducted in Women With Atopic Dermatitis Exposed to Ruxolitinib Cream Versus Topical Corticosteroids During Pregnancy: A US Claims Database Analysis — https://incyteclinicaltrials.com/studies/incb18424-ma-iai-403